CLINICAL TRIAL: NCT02661984
Title: A Randomized, Multi-Center, Single-Visit, Clinical Investigation to Assess the Degree of Agreement and Feasibility of Measuring Exhaled Nitric Oxide in Children, Aged 4-6 Years Old, With the NIOX VERO Using the 6 Second Exhalation Mode as Compared With the 10 Second Exhalation Mode
Brief Title: Measurement of FeNO in Young Children With the NIOX VERO
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Aerocrine AB (Industry)
Responsible Party: Sponsor
Other Study IDs: AER-052
Record Dates: First submitted 2016-01-05; First posted 2016-01-25 (Estimated); Last update posted 2017-05-15 (Actual); Status verified 2017-05

CONDITIONS: Asthma
Keywords: FeNO, exhaled nitric oxide
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Healthy (no pulmonary disease): Healthy children 4 - 6 years old with no pulmonary disease and not exhibiting respiratory illness or sinusitis.
- Asthmatic (physician diagnosed): Asthmatic children 4 - 6 years old not exhibiting acute asthma symptoms, respiratory illness or sinusitis.

SUMMARY:
FeNO measurements provide the physician with means of evaluating an asthma patient's response to anti-inflammatory therapy, as an adjunct to the established clinical and laboratory assessments in asthma. Interpretation of FeNO profiles is based on the nitric oxide plateau. To achieve plateau, the duration of exhalation must be sufficient (at least 4 seconds for children <12 years and > 6 seconds for children > 12 years (ATS/ERS, 2005).

Measurement of FeNO using the 6-sec mode may provide a viable alternative in children as young as age 4 years who may have difficulty maintaining exhalation for a full 10 seconds.

DETAILED DESCRIPTION:
The primary objective is to assess the degree of agreement of FeNO measured with the NIOX VERO using the 6-sec and 10-sec modes.

The secondary objectives of the Clinical Investigation are to:

* Assess the ability of participants to use the NIOX VERO for measuring FeNO in both exhalation modes, and
* Compare the repeatability of FeNO measured with the NIOX VERO in both exhalation modes.

Participants will attempt 2 measurements taken using the 6-sec mode followed by 2 measurements using the 10 second exhalation mode or vice versa.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female 4, 5 and 6 years old,
2. Primary Language: English or Spanish, and
3. Healthy (e.g., no pulmonary disease) or Asthmatic (if asthmatic, they must have a physician diagnosis of asthma).

Exclusion Criteria:

1. Pulmonary Disease Status: Any disease other than asthma.
2. In the opinion of the investigator, has severe or uncontrolled asthma (defined as having a) 2 or more exacerbations within the last year that required the use of systemic corticosteroids, or b) 1 or more hospitalizations, ICU stays or mechanical ventilations within the last year).
3. Has taken their reliever inhaler within 4 - 6 hours from the FeNO measurements.
4. Has acute asthma symptoms, respiratory illness (e.g. cold, flu), or sinusitis.
5. Has had food or beverage intake (other than water) or has participated in strenuous exercise within 1 hour prior to FeNO measurement.
6. Has a family relationship with the Operator or Study Personnel (persons who are family members of the Operator or Study Personnel are not eligible to participate).
7. Has a Parent/Guardian who is unable or unwilling to provide informed consent.

Ages: 4 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Healthy and Asthmatic 4 - 6 year old children.
Sampling Method: Non-Probability Sample
Enrollment: 102 (Actual)
Dates: Start 2016-01; Primary Completion 2016-11 (Actual); Study Completion 2017-05-31 (Estimated)

PRIMARY OUTCOMES:
The primary endpoint will be the analysis of the agreement of successful FeNO measurements in the 10 second and the 6 second exhalation modes. | After a single 1-2 hour visit
  This is a single visit study.

CONTACTS AND LOCATIONS:
Overall Officials: Kathy Rickard, MD, Study Director — Aerocrine AB
Locations (3):
- United States (3):
  - Arizona Allergy & Immunology Research, Gilbert, Arizona
  - Allergy and Asthma Specialists, Blue Bell, Pennsylvania
  - Allergy Partners of North Texas, Dallas, Texas

IPD SHARING:
Plan to Share IPD: No